CLINICAL TRIAL: NCT06559267
Title: School-based Paraeducator Education for Engagement at Recess
Acronym: SPEER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Freda Liu, Associate Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00020326; R324A240031 (Other Grant/Funding Number: Institute of Education Sciences)
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder; Neurodevelopmental Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: All schools that participate in the study will receive Remaking Recess. Additionally, half of the schools will be randomized to receive TEAM, an additional implementation support intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: (participants will be masked during randomization process, after randomization they will be informed which condition they receive. Outcomes assessors will be masked to randomization and randomization outcome to the best of our ability)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remaking Recess (Active Comparator): Remaking Recess is a school-based social engagement intervention designed to enhance elementary school contextual factors to better support peer engagement during recess. Remaking Recess is delivered to educators through direct training and in vivo coaching by a certified Remaking Recess Coach.
  Interventions: Behavioral: Remaking Recess
- TEAM (Experimental): Schools that are randomized to the TEAM condition will receive an additional implementation support intervention. TEAM will leverage existing human resources in the school to specifically focus on developing an implementation blueprint to foster a supportive implementation context for paraeducators to use Remaking Recess.
  Interventions: Behavioral: Remaking Recess; Other: TEAM

INTERVENTIONS:
Behavioral: Remaking Recess — Remaking Recess (RR) is a school-based social engagement intervention designed to enhance elementary school contextual factors to better support peer engagement during recess. Remaking Recess is delivered to educators through direct training and in vivo coaching by a certified Remaking Recess Coach.
  Other Names: RR
Other: TEAM — Schools that are randomized to the TEAM condition will receive an additional implementation support intervention. TEAM will leverage existing human resources in the school to specifically focus on developing an implementation blueprint to foster a supportive implementation context for paraeducators to use Remaking Recess.
  Other Names: TEAMS; school-based teams
  Arms: TEAM

SUMMARY:
The purpose of the proposed three-site study is to test whether an educator-level implementation strategy, coaching, with or without a school-level implementation strategy, school-based teams, will maximize paraeducators' use (fidelity and sustainment) of an evidence-based social engagement intervention, Remaking Recess (RR). RR aims to improve peer related social skills for autistic students and their non-autistic peers who are socially isolated or peripheral and need support during recess.

ELIGIBILITY:
Inclusion Criteria:

* Students: Elementary aged students in K-5th grade who are autistic or have a neurodevelopmental disorder (Age 5-12)
* Educators: Paraeducators, teachers, or other school personnel that work with K-5th grade students in a public school in the United States (Age 18+)

Exclusion Criteria:

* Students or educators that have previously participated in Remaking Recess studies will not be eligible to enroll in this study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Remaking Recess Fidelity | Baseline, 4 months, 8 months, 12 months, 16 months
  This 20-item observation measure rates how well educators are observed to be using core Remaking Recess strategies with students on the playground. Minimum score 1, maximum score 5. Higher scores indicate better outcome.

SECONDARY OUTCOMES:
Playground Observation of Peer Engagement (POPE) | Baseline, 4 months, 8 months, 12 months, 16 months
  This observation-based instrument measures children's engagement with activities and peers. It rates children's engagement states and the frequency within a set amount of time.
Friendship Survey | Baseline, 4 months, 8 months
  This 5-item free response survey asking students to identify their preferred peers at school. The results of the survey will be analyzed to identify student social network centrality in their classroom (Nuclear, Secondary, Peripheral, or Isolated).
Teacher Perceptions Measure | Baseline, 4 months, 8 months
  This 12-item measure asks teachers to report on their perceptions of their target student's social skills. Minimum score 1, maximum score 3. Higher scores indicate better outcome.
Acceptability of Intervention Measure (AIM) | Baseline, 4 months, 8 months, 12 months, 16 months
  This 12-item self-report measure asks educators to rate how acceptable the interventions (Remaking Recess and TEAM) were. Minimum score 1, maximum score 5. Higher scores indicate better outcome.
Cost Measure | Baseline, 4 months, 8 months, 12 months, 16 months
  This survey measure asks educators how much time they spent on study-related procedures (Remaking Recess and TEAM) each week. The measure then calculates the average dollar cost each week of study-related procedures based off of the educator's salary in order to better understand the cost of implementation and intervention.
Provider Report of Sustainment Scale (PRESS) | 12 months, 16 months
  This 3-item self-report measure asks educators to reflect on the sustainment of the use of the target intervention (Remaking Recess) at their school. Minimum score 0, maximum score 4. Higher scores indicate better outcome.
School Implementation Leadership Scale (S-ILS) | Baseline, 4 months, 8 months, 12 months, 16 months
  This 25-item measure captures educator perceptions of their school leadership and how well the leadership supports the use of the intervention (Remaking Recess). Minimum score 0, maximum score 4. Higher scores indicate better outcome.
School Implementation Climate Scale (SICS) | Baseline, 4 months, 8 months, 12 months, 16 months
  This 21-item measure captures educator perceptions of their school culture and how well the intervention (Remaking Recess) fits in. Minimum score 0, maximum score 4. Higher scores indicate better outcome.
Team Process Survey Measure (TPS) | Baseline, 4 months, 8 months, 12 months, 16 months
  A 10-item self-report measure to capture team process. Minimum score 1, maximum score 5. Higher scores indicate better outcome.
Quality of Play Questionnaire | Baseline, 4 months, 8 months, 12 months, 16 months
  A 19-item measure for parents/caregivers to complete about their child's playdates. Items 1-17 are a numerical rating of how much time a child spends on an activity in their play, with score ranging from a minimum of 0 to maximum of 3. Items 18-19 are a free response numerical frequency rating for parents to report on the number of playdates their child had in the last month.

CONTACTS AND LOCATIONS:
Overall Officials: Freda Liu, PhD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - University of California Los Angeles, Los Angeles, California
  - University of Oregon, Eugene, Oregon
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Locke J, Sridhar A, Shih W, Shire S, Eisman AB, Kim E, Du A, Espeland C, Kasari C. Study protocol for a hybrid type 3 effectiveness-implementation trial of a team-based implementation strategy to support educators' use of a social engagement intervention. Implement Sci. 2025 Jan 9;20(1):3. doi: 10.1186/s13012-024-01414-3. PMID 39789610